CLINICAL TRIAL: NCT02323009
Title: Esophageal Balloon Guided Weaning of the Morbidly Obese Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Minimal recruitment. very few patients available with eligibility criteria
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Ogugua N Obi, MD, MPH, Robert Shaw, MD (Principal Investigator), East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 10-0343
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Morbid Obesity
Keywords: Transpulmonary pressure; Esophageal balloon; Esophageal pressure monitoring device; Cstat; Static effective compliance; Ventilator weaning; Morbidly Obese Ventilator Dependent Tracheotomized Patients
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Esophageal balloon Arm (Active Comparator): Patients in this arm were randomly assigned to have their PEEP adjusted to maintain a positive transpulmonary pressure (0 to 10 cm H20).
  Interventions: Device: Esophageal Balloon
- Cstat Arm (Active Comparator): Patients in this arm had their PEEP adjusted to achieve the best static effective compliance (CStat).
  Interventions: Other: Cstat
- Historic Controls (No Intervention): These were historic controls with similar patient characteristics weaned by traditional methods in the 2-year period prior to the start of the study.

INTERVENTIONS:
Device: Esophageal Balloon — Esophageal balloon was used to measure esophageal pressure (Paux) which was used as an estimate of pleural pressure. Transpulmonary pressure (Ptp) was calculated as the difference between airway pressure (Pao) and Paux. Applied PEEP was then adjusted to overcome negative Ptp which we maintained between 0 to 10 cm H20. All measurements were made at end-expiration.
  Arms: Esophageal balloon Arm
Other: Cstat — PEEP was adjusted to achieve the best CStat in this group of patients
  Arms: Cstat Arm

SUMMARY:
This is a study to evaluate whether PEEP adjusted by use of an esophageal balloon to overcome negative transpulmonary pressure; or adjusted by use of "CStat" to achieve the best effective static compliance will have any effect on outcomes with respect to ventilator weaning in tracheotomized morbidly obese patients (BMI >=40) with at least one failed prior weaning attempt.

DETAILED DESCRIPTION:
Tracheotomized morbidly obese patients (BMI >= 40) who had failed an initial attempt at ventilator weaning (defined in the investigators study as ventilator dependent) were randomly assigned to one of two methods for setting Positive End Expiratory Pressure (PEEP).

Patients randomized to the esophageal balloon arm (ESO group) had their PEEP adjusted to overcome negative transpulmonary pressure and maintain a positive transpulmonary pressure (Ptp) of 0 to 10 cm H20 - targeting as close to zero as possible.

Patients randomized to the static effective compliance arm (CStat group) had their PEEP adjusted to achieve the best static effective compliance as automatically calculated and displayed on the graphic interphase of the hamilton G5 or Galileo ventilator. For this group, the PEEP was adjusted in increments of 3 cm H20 until there was a less than 5% observed improvement in the static effective compliance. the PEEP with the best Cstat was chosen.

At the end of the intervention period, this intervention cohort (termed "PEEP intervention cohort") will be compared to a group of historical controls to compare the efficiency of a PEEP-based weaning protocol to traditional weaning methods.

The investigators hypothesized that PEEP levels titrated by use of an esophageal balloon to maintain a positive transpulmonary pressure between 0 to 10 cm H20, would lead to improved outcomes with respect to ventilator weaning in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients with BMI of 40 or greater
* Ventilator dependent patients (defined as at least one prior failure at weaning)
* Tracheotomized
* No active underlying lung disease that would preclude ventilator weaning
* Stable hemodynamics
* Patient/ family able to give consent
* No naso-facial abnormalities that would interfere with placement of an esophageal balloon
* Fio2 <= 60%
* Patient able to tolerate Pressure Support ventilation

Exclusion Criteria:

* Lack of consent
* Patient deemed not weanable from mechanical ventilation as per the clinical judgement of the pulmonary physician
* Significant lung, heart or neuromuscular disease that would interfere with or preclude ventilator weaning, including an active ongoing lung infection.
* Contraindications to placement of an esophageal pressure monitoring device - such as ulcerations, tumors, diverticulitis, uncontrolled bleeding varices, sinusitis, epistaxis or recent nasopharyngeal surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of patients weaned by day 30 | 30-days
  A patient was considered successfully weaned and "ventilator independent" if they were spontaneously breathing without ventilator support for at least 24 hours, and remained off the ventilator by day 30. If ventilator support was subsequently required, the patient was returned to their original group and considered not weaned. The patients were considered to be weaned or not, after a period of thirty days.

SECONDARY OUTCOMES:
Time to wean | 30-days
  The time to wean/ time to achieve ventilator independence was measured from the date of randomization to the date of final successful liberation from mechanical ventilation. If patient had an unsuccessful initial wean, he was not considered weaned. Only patients who were considered weaned by day 30 accrued "time to ventilator independence."

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shaw, MD, Principal Investigator — East Carolina University
Locations (1):
- Vidant Medical Center, Greenville, North Carolina, United States

REFERENCES:
- [Background] Talmor D, Sarge T, O'Donnell CR, Ritz R, Malhotra A, Lisbon A, Loring SH. Esophageal and transpulmonary pressures in acute respiratory failure. Crit Care Med. 2006 May;34(5):1389-94. doi: 10.1097/01.CCM.0000215515.49001.A2. PMID 16540960
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Talmor DS, Fessler HE. Are esophageal pressure measurements important in clinical decision-making in mechanically ventilated patients? Respir Care. 2010 Feb;55(2):162-72; discussion 172-4. PMID 20105342
- [Background] Loring SH, Pecchiari M, Della Valle P, Monaco A, Gentile G, D'Angelo E. Maintaining end-expiratory transpulmonary pressure prevents worsening of ventilator-induced lung injury caused by chest wall constriction in surfactant-depleted rats. Crit Care Med. 2010 Dec;38(12):2358-64. doi: 10.1097/CCM.0b013e3181fa02b8. PMID 20890197
- [Background] Loring SH, O'Donnell CR, Behazin N, Malhotra A, Sarge T, Ritz R, Novack V, Talmor D. Esophageal pressures in acute lung injury: do they represent artifact or useful information about transpulmonary pressure, chest wall mechanics, and lung stress? J Appl Physiol (1985). 2010 Mar;108(3):515-22. doi: 10.1152/japplphysiol.00835.2009. Epub 2009 Dec 17. PMID 20019160
- [Background] Hedenstierna G. Esophageal pressure: benefit and limitations. Minerva Anestesiol. 2012 Aug;78(8):959-66. Epub 2012 Jun 14. PMID 22699701
- [Background] Owens RL, Campana LM, Hess L, Eckert DJ, Loring SH, Malhotra A. Sitting and supine esophageal pressures in overweight and obese subjects. Obesity (Silver Spring). 2012 Dec;20(12):2354-60. doi: 10.1038/oby.2012.120. Epub 2012 May 4. PMID 22695479
- [Background] MEAD J, GAENSLER EA. Esophageal and pleural pressures in man, upright and supine. J Appl Physiol. 1959 Jan;14(1):81-3. doi: 10.1152/jappl.1959.14.1.81. No abstract available. PMID 13630830
- [Background] Piraino T, Cook DJ. Optimal PEEP guided by esophageal balloon manometry. Respir Care. 2011 Apr;56(4):510-3. doi: 10.4187/respcare.00815. Epub 2011 Jan 21. PMID 21255501
- [Background] Washko GR, O'Donnell CR, Loring SH. Volume-related and volume-independent effects of posture on esophageal and transpulmonary pressures in healthy subjects. J Appl Physiol (1985). 2006 Mar;100(3):753-8. doi: 10.1152/japplphysiol.00697.2005. Epub 2005 Nov 23. PMID 16306256
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Derived] Obi ON, Mazer M, Bangley C, Kassabo Z, Saadah K, Trainor W, Stephens K, Rice PL, Shaw R. Obesity and Weaning from Mechanical Ventilation-An Exploratory Study. Clin Med Insights Circ Respir Pulm Med. 2018 Sep 18;12:1179548418801004. doi: 10.1177/1179548418801004. eCollection 2018. PMID 30245572